CLINICAL TRIAL: NCT04478617
Title: PROJECT PREVENT: Metronidazole Antibiotic Per Vagina Before Hysterectomy: Is Additional Antibiotic Prophylaxis Beneficial?
Acronym: PREVENT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14176
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Post-Op Infection
Keywords: Hysterectomy
MeSH Terms: interventions — Metronidazole; Benchmarking

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metronidazole (Experimental)
  Interventions: Drug: Metronidazole Vaginal
- Control (No Intervention)

INTERVENTIONS:
Drug: Metronidazole Vaginal — Vaginal metronidazole 0.75% (MetroGel or Vandazole) will be inserted per vagina days 1 through 5 prior to date of surgery.
  Other Names: MetroGel; Vandazole
  Arms: Metronidazole

SUMMARY:
Despite use of intravenous antibiotic prophylaxis, pelvic infection including vaginal and urinary complaints and infections are still noted after hysterectomy. For gynecologic surgery the burden of infection is not only from the skin but from the vagina and urinary tract. Hysterectomy involves a communication via the cervical or vaginal canal directly with the pelvis and thus can lead to a potentially increased risk of infection from both aerobic and anaerobic organisms. Vaginal metronidazole is a standard of care antibiotic for vaginal infections including bacterial vaginosis. Based upon small studies in the peri-operative setting, vaginal metronidazole may provide a benefit in decreasing surgical site infections and urinary infections in conjunction with standard infection prevention protocols.

This study is for women undergoing elective subtotal or total hysterectomy by any route of surgery. The main objective of this study is to evaluate if metronidazole inserted per vagina daily for 5 days before elective hysterectomy decreases patient complaints of potential infection or documented post-operative infection.

Subjects will be randomized to an intervention or control group. For subjects in the intervention group, vaginal metronidazole 0.75% (MetroGel or Vandazole) will be prescribed and inserted per vagina days 1 through 5 prior to date of surgery. The control group will not receive a metronidazole prescription.

DETAILED DESCRIPTION:
Standard of care surgical site infection (SSI) antibiotic prophylaxis for elective hysterectomy is a single intravenous antibiotic. Despite use of intravenous antibiotic prophylaxis, pelvic infection including vaginal and urinary complaints and infections are still often noted after hysterectomy. For gynecologic surgery the burden of infection is not only from the skin but from the vagina and urinary tract. Hysterectomy involves a communication via the cervical or vaginal canal directly with the pelvis and thus can lead to a potentially increased risk of infection from both aerobic and anaerobic organisms.

There has been scant retrospective data examining the use of metronidazole as an adjunct to standard antibiotic prophylaxis for hysterectomy. A few previous studies have examined the use of vaginal metronidazole in patients who had a documented overgrowth of normal bacterial flora (e.g. diagnosed with bacterial vaginosis) prior to hysterectomy in pre-menopausal women only and found a significant difference in prevention of infections.

Vaginal metronidazole is a standard of care antibiotic for vaginal infections including bacterial vaginosis. Based upon small studies in the peri-operative setting, vaginal metronidazole may provide a benefit in decreasing surgical site infections and urinary infections in conjunction with standard infection prevention protocols.

For post-operative patients, the symptoms of vaginal discharge, dysuria, pelvic pain and wound erythema/induration/drainage is not only distressing for the patient but leads to additional phone calls, patient visits, laboratory and radiology evaluation and possibly additional pain, and antibiotic prescriptions. This increased use of health care services can cause a burden to our health care system and diminish overall patient satisfaction. Therefore, if additional prophylaxis can also prevent patient reported symptoms of post-operative infection, the intervention may be of value.

The objective of this study is to investigate if metronidazole inserted per vagina daily for 5 days before elective hysterectomy decreases patient complaints of potential infection or documented post-operative infection.

Subjects randomized to the intervention are required to pick up the antibiotic at their own pharmacy. They must then insert the antibiotic per vagina once daily on days 1-5 (day 5 being the day before their scheduled operation).

There are no study related visits, imaging, or testing required above standard peri-operative procedures as per their gynecologic surgeon. Subjects randomized to the control group (no antibiotic) are followed for data collection only. Subjects in both groups will have a routine hospital stay for surgery and their routine follow up for post-operative care as per the standard practice of the gynecologic surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Any female aged 18 years old and over
* Patient scheduled for elective subtotal (removal of uterus only with or without ovaries) or total hysterectomy (removal of uterus and cervix with or without ovaries) by any route of surgery. Procedures will include laparoscopic, robotic, open and vaginal approaches.

Exclusion Criteria:

* Known hypersensitivity to metronidazole (oral or vaginal)
* Hysterectomy scheduled within 5 days of study enrollment (ie there will not be enough time to complete the study drug course)
* Suspected active bacterial vaginosis at time of consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Composite variable of patient reported symptom or documented post-operative infection by the 4 to 8-week post-operative visit(s). | 8 weeks following surgery.
  Patient reported symptom= patient report of dysuria, vaginal discharge with or without pelvic pain, fever, wound redness/erythema/drainage documented in the post-operative visit or complaint that generates an additional post-operative visit for evaluation.
  Documented post-operative infection= Urinary tract infection either empirically treated with antibiotics or culture proven infection, vaginal discharge with or without pelvic pain or that warrants treatment with antibiotics, vaginal cuff cellulitis or vaginitis, pelvic abscess (confirmed by pelvic ultrasound or CT scan with or without vaginal cultures) that results in antibiotic use.

SECONDARY OUTCOMES:
Individual rates of patient reported symptoms and documented post-operative infections by the 4 to 8-week post-operative visit. | 8 weeks following surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NYC Health + Hospitals/Metropolitan Hospital, New York, New York
  - Westchester Medical Center/New York Medical College, Valhalla, New York

REFERENCES:
- [Derived] Pradhan T, Zhang H, Kadesh A, Buskwofie A, Patankar S, Menon S, Ryntz T, Grimes CL. PROJECT PREVENT: a randomized controlled trial of preoperative vaginal metronidazole to decrease patient issues and infections after hysterectomy. BMJ Surg Interv Health Technol. 2024 Apr 4;6(1):e000241. doi: 10.1136/bmjsit-2023-000241. eCollection 2024. PMID 38596254